CLINICAL TRIAL: NCT03105206
Title: A Multicenter Prospective Research on the Treatment of Low Pole Renal Calculus by Flexible Ureteroscope
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Changzheng Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Tongji Hospital (Other); Renmin Hospital of Wuhan University (Other); The Second People's Hospital of GuangDong Province (Other); Jiangsu Provincial People's Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); West China Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng Gao, Changhai Hospital, Changhai Hospital
Other Study IDs: SHOT-20161208
Record Dates: First submitted 2017-04-02; First posted 2017-04-07 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Renal Calculus
Keywords: lowl pole renal calculus; anatomical parameters; flexible ureteroscopy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Low Pole Renal Calculus: patients with low pole renal calculus who are suitable to treat by flexible ureteroscopy
  Interventions: Procedure: Flexible Ureteroscopy

INTERVENTIONS:
Procedure: Flexible Ureteroscopy — the Treatment of Low Pole Renal Calculus by Flexible Ureteroscope

SUMMARY:
This study centers on the treatment of low pole renal stones by flexible ureteroscope and intends to find the key anatomical parameters using a prospective, randomized multi-center trial design and to make a more appropriate standard for flexible ureteroscopy of low pole renal stones.

DETAILED DESCRIPTION:
With the development of manufacturing technique, new generation of flexible ureteroscopes have great initiative and passive bending capacity and have greatly expanded its application. In our clinical practice, we have found that IPA (Infundibulopelvic angle) is no longer a decisive factor for the success of f-URS（flexible ureteroscope） surgeries. Thus, we think it is necessary to have further study on the effect of anatomy of renal collecting system for f-URS surgeries.

ELIGIBILITY:
Inclusion Criteria:

* • Subject has provided informed consent and indicated a willingness to comply with study treatments

  * Subject is 18-70 yrs of age
  * Subject can be either male or female
  * Subject has a diagnosis of low pole renal stones according to CT urography(CTU) or intravenous pyelogram (IVP) results
  * Subject has a single stone 1~2cm in size (KUB), or multiple stones 1~2cm in cumulative size (KUB), and is a surgical candidate for the ureteroscopic approach

Exclusion Criteria:

* • Subject has an active urinary tract infection (e.g., cystitis, prostatitis, urethritis, etc.)

  * Subject has been diagnosed with a urethral stricture or bladder neck contracture
  * Subject has been diagnosed with a urinary tract infection related to stone obstruction within two weeks
  * Subject has severe hematuria that might blur the vision of the endoscopy
  * Subject is pregnant or in monthly period
  * Subject has coexistent disease like systemic disease, heart disease, lung disfunction or other diseases that could not tolerate the endoscopic surgery or anesthesia.
  * Subject has unadjusted diabetes or high blood pressure
  * Subject has a disorder of the coagulation cascade system that would put the subject at risk for intraoperative or postoperative bleeding
  * Subject is unable to discontinue anticoagulant and antiplatelet therapy preoperatively (2 weeks)
  * Subject has been diagnosed with hydronephrosis larger than 3cm according to the B-scan ultrasonography examination
  * Subject has any kind of anatomic abnormality of the urinary system that might have an influence on the surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: low pole renal calculus patients
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
whether the f-URS could enter the low kidney calyx or not | during the operation
  Following conditions are regarded as failures: 1. the f-URS couldn't enter the low kidney calyx 2. Though the f-URS has entered the low kidney calyx, it cannot crush the stone.

SECONDARY OUTCOMES:
stone clearance | 4 weeks post-operatively
  Check NECT（nonenhanced CT）, no residual or residual stones are smaller than 2mm in total refers to clear success.Number of participants undergo f-URS surgeries without residual calculus/Total number of participants in each group *100%=stone clearance

CONTACTS AND LOCATIONS:
Overall Officials: Gao Xiaofeng, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Jessen JP, Honeck P, Knoll T, Wendt-Nordahl G. Flexible ureterorenoscopy for lower pole stones: influence of the collecting system's anatomy. J Endourol. 2014 Feb;28(2):146-51. doi: 10.1089/end.2013.0401. Epub 2013 Nov 19. PMID 24083332
- [Result] Resorlu B, Oguz U, Resorlu EB, Oztuna D, Unsal A. The impact of pelvicaliceal anatomy on the success of retrograde intrarenal surgery in patients with lower pole renal stones. Urology. 2012 Jan;79(1):61-6. doi: 10.1016/j.urology.2011.06.031. PMID 21855968
- [Result] Geavlete P, Jecu M, Geavlete B, Multescu R, Nita G, Georgescu D. Ureteroscopy--an essential modern approach in upper urinary tract diagnosis and treatment. J Med Life. 2010 Apr-Jun;3(2):193-9. PMID 20968209
- [Result] Madbouly K, Sheir KZ, Elsobky E. Impact of lower pole renal anatomy on stone clearance after shock wave lithotripsy: fact or fiction? J Urol. 2001 May;165(5):1415-8. PMID 11342888
- [Result] Lin CC, Hsu YS, Chen KK. Predictive factors of lower calyceal stone clearance after extracorporeal shockwave lithotripsy (ESWL): the impact of radiological anatomy. J Chin Med Assoc. 2008 Oct;71(10):496-501. doi: 10.1016/S1726-4901(08)70157-6. PMID 18955183
- [Result] Knoll T, Musial A, Trojan L, Ptashnyk T, Michel MS, Alken P, Kohrmann KU. Measurement of renal anatomy for prediction of lower-pole caliceal stone clearance: reproducibility of different parameters. J Endourol. 2003 Sep;17(7):447-51. doi: 10.1089/089277903769013577. PMID 14565873
- [Result] Wendt-Nordahl G, Mut T, Krombach P, Michel MS, Knoll T. Do new generation flexible ureterorenoscopes offer a higher treatment success than their predecessors? Urol Res. 2011 Jun;39(3):185-8. doi: 10.1007/s00240-010-0331-0. Epub 2010 Nov 5. PMID 21052986
- [Result] Geavlete P, Multescu R, Geavlete B. Pushing the boundaries of ureteroscopy: current status and future perspectives. Nat Rev Urol. 2014 Jul;11(7):373-82. doi: 10.1038/nrurol.2014.118. Epub 2014 Jun 3. PMID 24890883
- See also: Flexible ureterorenoscopy for lower pole stones: influence of the collecting system's anatomy — http://www.ncbi.nlm.nih.gov/pubmed/24083332
- See also: The impact of pelvicaliceal anatomy on the success of retrograde intrarenal surgery in patients with lower pole renal stones — http://www.ncbi.nlm.nih.gov/pubmed/21855968
- See also: Ureteroscopy--an essential modern approach in upper urinary tract diagnosis and treatment — http://www.ncbi.nlm.nih.gov/pubmed/20968209
- See also: Impact of lower pole renal anatomy on stone clearance after shock wave lithotripsy: fact or fiction — http://www.ncbi.nlm.nih.gov/pubmed/11342888
- See also: Predictive factors of lower calyceal stone clearance after extracorporeal shockwave lithotripsy (ESWL): the impact of radiological anatomy — http://www.ncbi.nlm.nih.gov/pubmed/18955183
- See also: Measurement of renal anatomy for prediction of lower-pole caliceal stone clearance: reproducibility of different parameters — http://www.ncbi.nlm.nih.gov/pubmed/14565873
- See also: Do new generation flexible ureterorenoscopes offer a higher treatment success than their predecessors? — http://www.ncbi.nlm.nih.gov/pubmed/21052986
- See also: Pushing the boundaries of ureteroscopy: current status and future perspectives — http://www.ncbi.nlm.nih.gov/pubmed/24890883